CLINICAL TRIAL: NCT02502370
Title: PRODIGE 33 - BALLAD - Phase III Trial Investigating the Potential Benefit of Adjvant Chemotherapy for Small Bowel Adenocarcinoma
Brief Title: Phase III Trial Investigating the Potential Benefit of Adjvant Chemotherapy for Small Bowel Adenocarcinoma
Acronym: BALLAD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: PRODIGE 33 - BALLAD
Record Dates: First submitted 2015-07-15; First posted 2015-07-20 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2015-07

CONDITIONS: Small Bowel Adenocarcinoma; Adjuvant Chemotherapy for SBA
MeSH Terms: interventions — Observation; Folfox protocol

ARMS (4):
- Group1 Arm A Observation (Active Comparator)
  Interventions: Drug: observation alone
- Group 1 Arm B LV5FU2 (Experimental)
  Interventions: Drug: LV5FU2
- Group 2 Arm C LV5FU2 (Active Comparator)
  Interventions: Drug: LV5FU2
- Group 2 ARM D FOLFOX (Experimental)
  Interventions: Drug: FOLFOX

INTERVENTIONS:
Drug: observation alone
  Arms: Group1 Arm A Observation
Drug: LV5FU2
  Arms: Group 1 Arm B LV5FU2; Group 2 Arm C LV5FU2
Drug: FOLFOX
  Arms: Group 2 ARM D FOLFOX

SUMMARY:
The utility of adjuvant chemotherapy in the management of Small Bowel Adenocarcinoma (SBA) remains unproven and awaits the results of a large, global, prospective, phase III, randomised, controlled trial. Across the 830 million population of North America and Europe, there are approximately 3,000 patients with stage I-III SBA every year who would be potentially eligible for such an adjuvant chemotherapy trial.

Given the absence of good-quality and evidence-based data, it has been agreed that a trial considering adjuvant chemotherapy versus no chemotherapy was appropriate for patients with stage I-III SBA in whom the oncologist and patient feel that the benefit of adjuvant chemotherapy is uncertain. For those patients with stage I-III SBA who, with their oncologists, feel that the potential benefit of adjuvant chemotherapy is certain (and hence are not willing to accept randomisation to the 'no chemotherapy' arm), a randomisation between single agent fluoropyrimidine versus doublet fluoropyrimidine and oxaliplatin chemotherapy will be offered. Tumour stage will be used as a stratification factor. Those patients who do not consent to be randomised will be offered registration to allow collection of demographic, clinicopathological and survival data, thereby making optimal use of the rare patient population available. In addition, archival Formalin Fixed Paraffin Embedded (FFPE) tissue and contemporaneous venous blood samples will be collected from every registered patient to allow molecular profiling and future translational research. A questionnaire about underlying risk factors (e.g. Crohn's disease, coeliac disease, Lynch syndrome etc) will be completed along with the other collected data on all registered patients.

ELIGIBILITY:
Inclusion Criteria:

1. R0 resected stage I, II or III small bowel adenocarcinoma
2. No evidence of residual or metastatic disease at laparotomy and CT/MRI imaging of chest, abdomen and pelvis.
3. Patients must be registered and randomised within 12 weeks of surgery and commence chemotherapy within 14 weeks of surgery
4. ECOG Performance Status of 0 or 1
5. Absolute neutrophil account ≥ 1.5 x109/l
6. Platelet count ≥ 100 x 109/l
7. Haemoglobin ≥90 g/l (previous transfusion is allowed)
8. AST and ALT ≤ 2.5 x upper limit of normal (ULN). (At least one of ALT or AST MUST be performed)
9. Creatinine clearance > 50 ml/min (calculated by Cockcroft Gault or Wright equation) or measured by EDTA
10. Serum bilirubin ≤ 1.5 x ULN
11. Signed and dated informed consent indicating that the patient has been informed of all the pertinent aspects of the trial prior to enrolment.
12. Age ≥ 16 years
13. Willingness and ability to comply with scheduled visits, treatment plans and laboratory tests and other trial procedures.

Exclusion Criteria:

1. Non-adenocarcinoma histology of small bowel tumour which includes but is not confined to lymphoma, GIST, carcinoid or other neuroendocrine tumour, squamous carcinoma, melanoma or sarcoma.
2. Previous neo-adjuvant chemo(radio)therapy for small bowel adenocarcinoma
3. Clinically significant cardiovascular disease (i.e. active or < 12 months since cerebrovascular accident, myocardial infarction, unstable angina, New York Heart Association [NYHA] grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, uncontrolled hypertension)
4. Pregnancy/lactation or of child bearing potential and not using medically approved contraception. (Postmenopausal women must have been amenorrhoeic for at least 12 months to be considered of non-childbearing potential)
5. Previous malignancy other than adequately treated in situ carcinoma of the uterine cervix or basal or squamous cell carcinoma of the skin, unless there has been a disease free interval of at least 3 years and treatment was with curative intent
6. Known or suspected dihydropyrimidine dehydrogenase (DPD) deficiency
7. Known untreated coeliac disease (may be enrolled if diet controlled), untreated chronic inflammatory bowel disease or other cause of malabsorption or intestinal obstruction
8. Grade ≥ 2 peripheral neuropathy
9. Administration of any investigational drug within 28 days or 5 half-lives, whichever is longer, prior to receiving the first dose of trial treatment.
10. Previous hypersensitivity to platinum salts
11. Patients with clinically significant active infections, or any other serious medical condition in which chemotherapy is contraindicated will be excluded
12. Patients with untreated vitamin B12 deficiency are excluded from receiving folinic acid as part of their chemotherapy regimen. However, these patients may be eligible for treatment with capecitabine fluoropyrimidine therapy, where no folinic acid is administered as part of the treatment regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Primary Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
The 3-year disease-free survival | 3 years
Overall survival | 7 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU du Bocage, Dijon, France

REFERENCES:
- [Derived] Kitahara H, Honma Y, Ueno M, Kanemitsu Y, Ohkawa S, Mizusawa J, Furuse J, Shimada Y; Colorectal Cancer Study Group and Hepatobiliary and Pancreatic Oncology Group of the Japan Clinical Oncology Group. Randomized phase III trial of post-operative chemotherapy for patients with stage I/II/III small bowel adenocarcinoma (JCOG1502C, J-BALLAD). Jpn J Clin Oncol. 2019 Mar 1;49(3):287-290. doi: 10.1093/jjco/hyy188. PMID 30590606